CLINICAL TRIAL: NCT02401139
Title: Ketamine Therapy Among Patients With Treatment-resistant Depression: a Randomised, Double-blind, Placebo-controlled Trial: Pilot Phase
Brief Title: Ketamine Trial for the Treatment of Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Principal Investigator, Colleen Loo, Professor, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HREC 15009
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2023-03-30 (Actual); Status verified 2015-03

CONDITIONS: Unipolar Depression
MeSH Terms: conditions — Depressive Disorder | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment arm (Active Comparator): Ketamine
  Interventions: Drug: Ketamine
- Placebo arm (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine
  Arms: Treatment arm
Drug: Placebo
  Arms: Placebo arm

SUMMARY:
This study is a Randomized Controlled Trial, investigating the safety and efficacy of administration of ketamine as a potential treatment for depression.

ELIGIBILITY:
Individuals will be eligible for enrolment on the basis of:

* major depressive disorder for at least three months duration
* an inadequate response to at least 2 adequate antidepressants
* MADRS ≥ 20

Patients will be excluded on the basis of:

* History of psychosis
* History of bipolar disorder
* Any unstable medical or neurologic condition
* Any Axis I disorder other than MDD judged to be primary presenting problem
* Planned major changes to psychotropic medication
* Significant risk of suicide
* Planned or probable use of ECT
* Age under 16 years, or 16-17 years without parental consent
* Substance abuse or dependence in previous 6 months
* Any history of abuse of ketamine or phencyclidine
* Contraindication to the use of ketamine
* Planned use of ketamine
* Women of childbearing potential not taking reliable contraception
* Likely non-compliance with trial treatment
* Other condition judged by the treating clinician as likely to impact on the ability of the participant to complete the trial

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale for Depression (MADRS) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Colleen K Loo, MBBS, MD, Principal Investigator — University of New South Wales
Locations (2):
- Australia (2):
  - Brain & Mind Research Institute (BMRI), University of Sydney, Camperdown, New South Wales
  - Black Dog Institute, University of New South Wales, Sydney, New South Wales